CLINICAL TRIAL: NCT02929303
Title: Expanded Access of Omegaven IV Fat Emulsion (Fish Oil Infusion) to Infants and Children With Parenteral Nutrition-associated Liver Disease
Brief Title: Expanded Access of Omegaven IV Fat Emulsion to Infants and Children With PNALD
Status: Approved for marketing | Type: Expanded Access
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: K5900315
Record Dates: First submitted 2016-09-13; First posted 2016-10-11 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis

INTERVENTIONS:
Drug: Omegaven IV lipid emulsion — Therapy is started at a dose of 1 gm/kg/day over 12 hrs. Omegaven may be infused via a central or peripheral IV. If additional fat calories are needed they will be provided by the enteral route.

SUMMARY:
This is an expanded access protocol for use of intravenous fish oil infusion, Omegaven, in infants and children with parenteral nutrition associated liver disease (PNALD) to decrease elevated liver enzymes and direct bilirubin.

This study aims to describe the response of PNALD after use of Omegaven by normalization of serum levels of liver enzymes and bilirubin.

DETAILED DESCRIPTION:
The etiology of parenteral nutrition associated liver disease (PNALD) is currently considered multifactorial. Available treatment options for this disease process are limited and have achieved moderate success at best. Unlike conventional intravenous fat emulsions, Omegaven™ is comprised solely of fish oils containing primarily omega-3 fatty acids. The investigators hypothesize that administering Omegaven™ to patients with PNALD in place of conventional fat emulsion may reverse cholestasis allowing patients to be maintained on adequate PN until they are able to ingest adequate nutrition enterally.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aged 0 - 18 yrs
2. Patients will be PN dependent (unable to meet nutritional needs solely by enteral nutrition). It will be assumed that patients will require parenteral nutrition for at least 30 days from the inclusion into the study.
3. Patients must have parenteral nutrition associated liver disease (PNALD) as defined as a direct bilirubin of 2mg/dl or more. Other causes of liver disease should be excluded. A liver biopsy is not necessary for treatment.
4. 2 consecutive direct bilirubins > 2.0 mg/dl. one week apart.
5. Signed patient informed consent.
6. The patient must have utilized standard therapies as clinically appropriate to prevent the progression of his/her liver disease. Such therapies could include surgical treatment, cyclic PN, avoiding overfeeding, reduction/removal of copper and manganese from PN, advancement of enteral feeding, and the use of ursodiol (i.e.,Actigall).

Exclusion Criteria:

1. Documented cause of chronic liver disease other than parenteral nutrition associated liver disease.
2. An allergy to any seafood product, egg protein, and/or previous allergy to Omegaven.
3. Active coagulopathy characterized by ongoing bleeding or by a requirement for clotting factor replacement (e.g. fresh frozen plasma or cryoprecipitate) to maintain homeostasis.
4. Impaired lipid metabolism or severe hyperlipidemia with or without pancreatitis.(e.g. (triglycerides > 1000mg/dl while receiving intralipid 1g/kg/day or less)
5. Unstable diabetes mellitus or hyperglycemia (Blood glucose >200 mg/dL) at the time of initiation of Omegaven
6. Currently being treated for stroke, embolism, collapse and shock, myocardial infarction.
7. Cholestasis due to any reason other than parenteral associated liver disease
8. Active new infection at time of initiation of Omegaven
9. Hemodynamic instability (e.g. receiving vasopressors) at time of initiation of Omegaven.
10. The patient may not be enrolled in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team).
11. Known pregnancy.

Max Age: 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Hector Hernandez, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Children's Hospital, Park Ridge, Illinois, United States

REFERENCES:
- [Result] Sant'Anna AM, Altamimi E, Clause RF, Saab J, Mileski H, Cameron B, Fitzgerald P, Sant'Anna GM. Implementation of a multidisciplinary team approach and fish oil emulsion administration in the management of infants with short bowel syndrome and parenteral nutrition-associated liver disease. Can J Gastroenterol. 2012 May;26(5):277-80. doi: 10.1155/2012/571829. PMID 22590701
- [Result] Soden JS, Lovell MA, Brown K, Partrick DA, Sokol RJ. Failure of resolution of portal fibrosis during omega-3 fatty acid lipid emulsion therapy in two patients with irreversible intestinal failure. J Pediatr. 2010 Feb;156(2):327-31. doi: 10.1016/j.jpeds.2009.08.033. PMID 20105644